#### NCT# 00911079

# UNIVERSITY OF CALIFORNIA, SAN FRANCISCO CONSENT TO PARTICIPATE IN A RESEARCH STUDY

Study Title: CC#08992: A Pilot Study of Catheter-Based Ultrasound Hyperthermia System

This is a clinical trial, a type of research study. Your study doctors, I-Chow Hsu, M.D., and Chris Diederich, PhD, from the UCSF Department of Radiation Oncology, will explain the clinical trial to you.

Clinical trials include only people who choose to take part. Please take your time to make your decision about participating. You may discuss your decision with your family and friends and with your health care team. If you have any questions, you may ask your study doctor. The National Cancer Institute (NCI) booklet, "Taking Part in Cancer Research Treatment Studies", is also available from your doctor.

You are being asked to take part in this study because you have advanced or recurrent cancer located in your pelvic region (cervix, uterus, prostate) and part of your cancer treatment requires temporary internal radiation treatments (also called radiotherapy or brachytherapy) which involves temporarily placing a radioactive source inside a thin flexible tube (catheter) near your tumor to deliver radiation to the tumor.

## Why is this study being done?

This study will use a device called an ultrasound applicator that creates heat using sound waves that cannot be heard by the human ear. The ultrasound devices fit inside the catheters used for your brachytherapy and are used to increase the tumor's temperature. Treatment with heat is called hyperthermia treatment. The purpose of this study is to find out whether the temperatures that we believe are effective can be reached using this device and to learn if hyperthermia can be done safely and appropriately using this device. The device is considered investigational by the FDA and has not been approved for use outside of this study.

This study is sponsored by the National Institutes of Health.

## How many people will take part in this study?

24 people will take part in this study.

### What will happen if I take part in this research study?

If you take part in this study, in addition to your brachytherapy treatments, you will receive two hyperthermia treatments, one during each two of your brachytherapy sessions.

## Before you begin the study...

A medical history and physical examination will be done by the doctor who will perform the brachytherapy.

IRB NUMBER: 10-03844 IRB APPROVAL DATE: 07/25/2019 sity of California IRB EXPIRATION DATE: 07/24/2020

## During the study...

## Brachytherapy (internal radiation therapy)

Brachytherapy is a standard part of your radiation treatment for your cancer. As part of your treatment you may also receive x-ray therapy and chemotherapy. Brachytherapy involves the insertion of catheters (small plastic tubes), so the radioactive source may be temporarily placed inside them to deliver radiation to the tumor. This is called an implant session. The catheters are inserted in the operating room, while you are under general anesthesia. General anesthesia puts you to sleep so you won't feel or remember surgical procedures.

After the catheters are inserted, a CT or MRI scan of the implanted catheters is done. Information from the scan will help the physician to plan the brachytherapy and hyperthermia. A typical brachytherapy treatment takes 5-30 minutes. You will receive a total of 2-3 treatments over 24 hours with each implant session (hospital stay). Each treatment will be given in a special treatment room. You will not be radioactive when the treatment is finished. After the last treatment of the implant session is completed, the catheters will be removed before you are discharged.

For the MRI test, you may receive gadolinium (a contrast agent) through a vein in your arm. Gadolinium is an agent that causes some tumors to appear much brighter than normal tissue on MRI scans; before gadolinium is injected the tumor may not be visible. A tiny tube inserted into a vein may be placed in your arm to inject the contrast agent. You will then lie down on a narrow bed which will be placed in a tunnel that is 6 feet long by 2 feet wide and open at each end. You will lie there quietly for about one hour, during which time you will hear a loud machine-like noise. The MRI scan is done in the radiology department and takes approximately 1.5 hours.

A CT scan is a special type of x-ray that allows your doctors to create a picture of the inside of your body in order to determine the size and location of your cancer. For the CT scan, you will receive a "contrast agent" - this is a special dye that is used to get clearer pictures of your body cavity. The contrast agent will be given to you through a needle in a vein in your arm. You will lie flat on a table that will move you into the CT scan machine. You will be asked not to move and may be asked to hold your breath for a few seconds periodically. The CT scan takes approximately 30 minutes.

### **Hyperthermia**

The purpose of hyperthermia is to enhance the effect of radiotherapy (brachytherapy) by increasing the tumor temperature to about 109°F, for about 60 minutes. The increase in temperature is achieved using special ultrasound applicators. The ultrasound applicators are designed to fit in the brachytherapy catheters. During treatment, you may feel warmth near the catheter.

To measure the heat created by the ultrasound, temperature probes will be placed in some of the catheters. Additional temperature probes will be placed in other catheters that are inserted in the bladder and rectum to monitor temperature. Tissue temperature around the applicator will be monitored continuously during the hyperthermia. However, if you feel the temperature is too hot or cannot tolerate the treatment for any reason, then the applicator power may be turned down or the hyperthermia treatment stopped by removing the applicator.

IRB NUMBER: 10-03844 IRB APPROVAL DATE: 07/25/2019 IRB EXPIRATION DATE: 07/24/2020

CC# 08992

During your first and second implant sessions, hyperthermia is given within 1 or 2 hours after one of the brachytherapy treatments in each implant session. If your doctor decides you need more than two implant sessions, only brachytherapy will be done, and hyperthermia will not be done

#### When I am finished with the treatment...

You will have follow-up visits with your study doctor at 1 month and at 3 months after completion of the treatment. Information collected at these routine visits will be used for study purposes. If you think you are having side effects from the treatment before it is time for your 1 month followup visit, it is important that you tell your study doctor, I-Chow Hsu. You can tell the doctor in person or call him

## How long will I be in the study?

The typical brachytherapy implant session (insertion of the catheters near the tumor site and treatment with radiation) requires a 1-night hospital stay, where you will receive 2-3 brachytherapy treatments over 24 hours. The first hyperthermia treatment will be done shortly after one of the brachytherapy treatments of the first implant session. The second brachytherapy implant session will be done after 1 to 3 weeks, and the second hyperthermia treatment will be done after a brachytherapy treatment during the second implant session. Since the hyperthermia is delivered during the same hospital stay as your brachytherapy treatments, it will not prolong your hospital stay. If your doctor decides you need additional brachytherapy sessions, you will not have hyperthermia again after the second session. Followup visits will be scheduled at 1 month and 3 months after the completion of hyperthermia treatment. These visits will take less than 1 hour.

## **Study Plan**

Another way to find out what will happen to you during the study is to read the chart below. Start reading at the top and read down the list, following the arrows. Only the parts that are **bolded** and underlined are being done as part of the study; the other parts would be done as part of your regular brachytherapy treatment even if you choose not to take part in the study.

> Physical Exam and Medical History before brachytherapy treatment Hospital admission for first brachytherapy implant session

Brachytherapy catheters implanted (Implant Session #1)

MRI or CT

Brachytherapy treatments using Session #1 catheter implants on the same day and/or the next day - **Ultrasound Hyperthermia** will follow one of these brachytherapy treatments

> Removal of session #1 catheters Hospital discharge



Brachytherapy treatments using Session #2 catheter implants on the same day and/or the next day - <u>Ultrasound Hyperthermia</u> will follow one of these brachytherapy treatments (this is the last hyperthermia treatment)

If medically necessary, additional Brachytherapy implant sessions (without Ultrasound Hyperthermia treatment)

# 1-month and 3-month study follow-up

## Can I stop being on the study?

Yes. You can decide to stop at any time. Tell the study doctor if you are thinking about stopping or decide to stop.

The researcher may decide to take you off this study if it is in your best medical interest, your condition worsens, or new information becomes available and this information suggests that the treatment will be ineffective or unsafe for you. It is unlikely, but the study may be dropped due to lack of funding or participation. You can stop participating at any time. However, if you decide to stop participating in the study, we encourage you to talk to the researcher and your regular doctor first.

## What side effects or risks can I expect from being in the study?

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop the treatment. In some cases, side effects can be serious, long lasting, or may never go away. You should talk to your study doctor about any side effects that you have while taking part in the study.

Risks and side effects related to HDR brachytherapy and heating tissue with ultrasound during hyperthermia treatment include those which are:

### Likely (>50% of subjects)

- Soreness in treated area
- Fatique
- Bowel irritation with increased frequency and urgency

Less Likely (>10-50% of subjects)

- Bladder irritation with increased feelings of needing to urinate and possibly feeling like you need to urinate suddenly
- Vaginal narrowing and shortening
- Painful intercourse
- Nausea
- Heat damage to healthy tissue
- Pain
- Irritation of skin or other soft tissue
- Blister(s)

#### Rare but serious (1-10% of subjects)

- Bleeding
- Open sores
- Blockage in the bowel
- Abnormal opening between bladder/vagina
- Abnormal opening between rectum/vagina
- Abnormal opening between rectum/prostate
- Infection
- Formation of scar tissue causing firm or thickened tissue in the area of brachytherapy
- Death of healthy tissue surrounding the tumor area
- Serious complication including death from anesthesia (<1%)</li>

Risks related to the other procedures being done in this study include:

#### CT scan risks

CT scans will expose you to controlled amounts of radiation. Although in theory any amount of radiation can be harmful, the total dose of radiation from these tests will be small and should not harm you. Some people may experience feelings of anxiety or claustrophobia while undergoing a CT scan.

#### MRI scan risks

The MRI machine acts like a giant magnet, and precautions will be taken so that loose metal objects do not move around the room and harm you. Things such as pocketknives or keychains are not allowed in the MRI room, and if you have a piece of metal in your body (such as ear implants, a pacemaker, or aneurysm clips) you will not be allowed in the MRI room. The MRI machine also makes a loud banging noise which has caused temporary hearing loss in some patients, so you will be asked to wear earplugs. You may also feel warm during the scan. You will be asked to remain still and not swallow for a while, which can be uncomfortable. Some people may experience feelings of anxiety or claustrophobia while undergoing an MRI scan.

#### Contrast material/Dye risks

The CT scans and MRI scans may require that a dye (contrast material) be injected into your vein through an intravenous (i.v.) line. There is a risk of an allergic reaction to the dye, although this is rare. Allergic reactions may include nausea, flushing, a 'pins and needles' sensation, mild headache, skin rash, itchy eyes, shortness of breath, and lightheadedness or low blood pressure (which can be treated with intravenous fluids).

In rare cases, the contrast material used for CT scans may cause injury to your kidneys. This is more likely to happen in patients with preexisting kidney problems.

IRB NUMBER: 10-03844 IRB APPROVAL DATE: 07/25/2019 ity of California IRB EXPIRATION DATE: 07/24/2020

#### Gadolinium risks

Patients with severe kidney disease sometimes have a bad reaction to gadolinium contrast. The condition is called nephrogenic sclerosing fibrosis (NSF). It can cause skin to tighten or scar and can damage internal organs. Sometimes it can be life-threatening. There are no reports of NSF in patients with normal kidney function. Before you have an MRI requiring an injection of gadolinium contrast, you will have a blood test in order to check the function of your kidneys. Based on your medical history and the results of the test, a doctor will decide whether it is safe for you to undergo the MRI.

## Are there benefits to taking part in the study?

Taking part in this study may or may not make your health better. While doctors hope that heating tumor tissue using Ultrasound Hyperthermia after Brachytherapy will be more useful against cancer compared to Brachytherapy alone, there is no proof of this yet. Other studies combining hyperthermia with radiation therapy and chemo-radiation therapy for cancer have shown significant improvements in response and survival. We hope the information learned from this study will benefit other patients with similar cancer in the future.

## What other choices do I have if I do not take part in this study?

Your other choices may include:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting no treatment
- Referral to another institution delivering hyperthermia
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible

Talk to your doctor about your choices before you decide if you will take part in this study.

#### Will my medical information be kept private?

We will do our best to keep your personal information confidential. We cannot guarantee absolute confidentiality. No individual identifiers will be used in any reports or publications resulting from this study, but the data will be used in the interests of the research ongoing at this center. Records of your progress while on the study will be kept in confidential form at this institution. Your personal information may be disclosed if required by law.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The National Cancer Institute (NCI) and other government agencies, e.g., the Food and Drug Administration (FDA), involved in keeping research safe for people.
- The University of California

Participation in research may involve a loss of privacy, but information about you will be handled as confidentially as possible. A medical record will be created because of your participation in this study. Your consent form and some of your research test results will be included in this record. Therefore, your other doctors may become aware of your participation. Hospital regulations require that all health care providers treat information in medical records confidentially.

IRB NUMBER: 10-03844 IRB APPROVAL DATE: 07/25/2019 ty of California IRB EXPIRATION DATE: 07/24/2020

#### What are the costs?

You and/or your health plan/health insurance company will need to pay for some or all of the costs of treating your cancer. Taking part in this study is not likely to cost you or your insurance company more than the cost of getting regular cancer treatment.

You will not be charged for the experimental ultrasound hyperthermia treatment. Only your standard cancer treatments will be charged to you or your health insurance.

For more information on clinical trials and insurance coverage, you can visit the National Cancer institute's web site at http://cancer.gov/clinicaltrials/understanding/insurance-coverage. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

## Will I be paid for taking part in this study?

You will not be paid for taking part in this study.

## What happens if I am injured because I took part in this study?

It is important that you tell your study doctor, I-Chow Hsu, M.D., if you feel that you have been injured because of taking part in this study. You can tell the doctor in person or call him

Treatment and Compensation for Injury: If you are injured as a result of being in this study, treatment will be available. The costs of the treatment may be covered by the University of California, depending on a number of factors. The University does not normally provide any other form of compensation for injury. For further information about this, you may call the office of the Committee on Human Research at (415) 476-1814.

### What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek compensation by signing this form.

#### Who can answer my questions about the study?

You can talk to your study doctor about any questions, concerns, or complaints you have about this study. Contact your study doctor, I-Chow Hsu, M.D.

If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you mayhave about the study, please call the Office of the Committee on Human Research at (415) 476-1814.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### CONSENT

You have been given copies of this consent form and the Experimental Subject's Bill of Rights to keep.

You will be asked to sign a separate form authorizing access, use, creation, or disclosure of health information about you.

PARTICIPATION IN RESEARCH IS VOLUNTARY. You have the right to decline to participate or to withdraw from this study at any time without penalty or loss of benefits to which you are otherwise entitled.

If you wish to participate in this study, you should sign below.

| Participant's i | name (PRINT) |
|---|---|
| Date | Participant's Signature for Consent |
| Date | Signature of Person Obtaining Consent |
| Date | Signature of Witness (Only required if the participant is a non-English speaker) |